CLINICAL TRIAL: NCT00694122
Title: Comparison of Lantus and NPH Insulin in the Dawn Phenomenon
Brief Title: Comparison of Lantus and Neutral Protamine Hagedorn (NPH) Insulin in the Dawn Phenomenon
Acronym: DAWN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, David M. Nathan, MD, Director, Diabetes Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-P-002515/24
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes; Dawn Phenomenon
Keywords: glucose; cortisol; growth hormone; glucagon; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glargine (Lantus) insulin (Active Comparator): Long acting insulin, glargine, that subject currently used as an outpatient. SC injections. Dose given at 22:00 is based on past week blood glucose data during evening overnight hours and AM glucose. 20.2 +/- 11.7 units glargine (mean +/- SD).
  Glargine (Lantus): Sanolfi Aventis
  Hourly blood glucose from 22:00 to 08:00 while receiving glargine (Lantus) insulin will be compared with the NPH insulin arm.
  Interventions: Drug: Lantus (glargine)
- NPH insulin (Active Comparator): Long acting insulin, NPH, that participant was currently while an outpatient. SC injections. Dose (units) given at 22:00 is based on past week blood glucose during evening overnight period and AM glucose. 20.7 +/- 10.0 units NPH (mean +/- SD).
  NPH: Eli Lilly
  Hourly blood glucose from 22:00 to 08:00 while receiving glargine (Lantus) insulin will be compared with the glargine (Lantus) insulin arm.
  Interventions: Drug: Lantus (glargine)

INTERVENTIONS:
Drug: Lantus (glargine) — Described in Arm Description
  Other Names: Lantus (glargine): Sanolfi Aventis; NPH: Eli Lilly

SUMMARY:
1. To investigate the effect of insulin glargine (Lantus™) vs NPH insulin regarding glycemic control during the early AM (dawn phenomenon) in individuals with type 1 diabetes.
2. To measure hormones implicated in the pathogenesis of the dawn phenomenon in individuals with type 1 diabetes.

DETAILED DESCRIPTION:
Title: COMPARISON of LANTUS and NPH INSULIN IN THE DAWN PHENOMENON

I. Background and Significance

Diabetes mellitus affects greater than 6% of the population, with type 2 more prevalent than type 1. For individuals with type 1 diabetes, the challenge has been to replicate insulin secretion of the healthy pancreas to maintain blood glucose as close to the non-diabetic range as possible. Insulin regimes using insulins with varied activity profiles (multiple daily injections or MDI) and continuous subcutaneous insulin infusion (CSII) have been somewhat successful in "mimicking" normal pancreatic function (1, 2). For individuals with type 1 diabetes, the benefits of near-normal, long-term glycemic control in delaying the development and slowing the progression of long-term complications was demonstrated in the Diabetes Control and Complications Trial (3). Intensive insulin therapy to achieve near-normal glycemic control has been limited by a three-fold increase in episodes of hypoglycemia (3, 4). Insulin analogs that provide more stable physiologic insulin levels have led to the development of newer MDI regimes (5). Glargine (Lantus) is a long-acting recombinant human insulin analog demonstrated to provide a continuous, smooth supply of insulin with no pronounced peak over a 24-hour period (6).

An increase in blood glucose in type 1 and type 2 diabetics, and an increase in insulin secretion to maintain normoglycemia in non-diabetics, was documented in several studies in the 1980s (15-17). This physiological requirement for more insulin delivery (or secretion) in the early (4:00-6:00 AM) hours was termed the "dawn phenomenon". The mechanism for the dawn phenomenon was thought to be the overnight increase in growth hormone section, rather than diurnal glucocorticoids (16, 18, 19). Most intensive treatment regimens of the 1980-90's, with MDI or CSII, were designed to provide more insulin in the 4:00-7:00 AM period to cope with the dawn phenomenon which cannot be be achieved with glargine (20-21). Continuous monitoring of blood glucose has revealed that individuals treated with CSII had significantly better glycemic control than glargine treated individuals (22). Whether the dawn phenomenon, with increased area under the curve blood glucose levels during the dawn period is limiting the effectiveness of regimens with glargine is of crucial importance.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to performing screening evaluations.
* Male or female, 18 yrs or older.
* Diagnosis of type 1 diabetes made 5 years prior to screening visit.
* A1C > 6.0% and 9.0% at screening visit.
* Body Mass Index (BMI) 35 kg/m2 at screening visit.
* Documented undetectable C-Peptide
* Ability to follow instructions for Continuous Glucose Monitoring System (CGMS).
* Multiple daily injection participants on at least 3 injections per day. May be treated with NPH or glargine.

Exclusion Criteria:

* Pregnant or lactating females, or females planning to become pregnant during the study or not using an acceptable method of contraception. Females of childbearing potential must have a negative pregnancy test at Visit 3 and Visit 5. Females who become pregnant during the study will be discontinued.
* Type 2 diabetes.
* Two or more severe hypoglycemic episodes (requiring assistance) within six months of Screening.
* Drugs known to affect glycemia (eg. steroids, beta blockers) or conditions that are likely to require steroid therapy or cause metabolic instability in the next 6 months.
* History of allergy or intolerance to NPH or glargine.
* History of hypoglycemia unawareness i.e. no warning symptoms accompanying low (<50 mg/dl) blood glucose levels.
* Unable and/or unlikely to comprehend and/or follow the study protocol (including self blood glucose monitoring, CGMS).
* Currently using an insulin pump.
* Pituitary disorder (Acromegaly, Cushing's, Hypothyroidism etc.) or tumor.
* Two or more severe hypoglycemic episodes (requiring assistance) within six months of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Nathan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusettes General Hospital/ Diabetes Research Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January 2007 and ended on January 2011. Individuals were recruited from the MGH Diabetes Center, MGH internal Research Broadcast for research volunteers. Advertisements were placed in the local metro and flyers posted around the institution, altho no participants contacted study staff from these latter advertisemens.
Pre-assignment Details: 200 participants were recruited; 43 were phone screened; 27 signed consent forms, 12 exluded (3 did not meet inclusion criteria, 7 no longer wanted to participate and 3 lost to follow-up).
Groups:
- Lantus First, Then NPH: Lantus insulin once per day and blood glucose outcomes was studied during the first overnight visit; then the subject was discharged on NPH on twice per day NPH. Upon the second overnight visit, NPH insulin and blood glucose outcomes was studied
- NPH First, Then Lantus: NPH was given twice per day in the first intervention period for 3-4 weeks and .Lantus was given once per day in second intervention period for 3-4 weeks.
Period: First Intervention (3-4 Weeks)
Arm/Group | Lantus First, Then NPH | NPH First, Then Lantus
Started | 20 (Started Lantus then on NPH.) | 7 (Started on NPH then on Lantus.)
Completed | 10 | 5
Not Completed | 10 | 2
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Did not meet entrance criteria | 2 | 1
Period: Washout (1 Day)
Arm/Group | Lantus First, Then NPH | NPH First, Then Lantus
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0
Period: Second Intervention (3-4 Weeks)
Arm/Group | Lantus First, Then NPH | NPH First, Then Lantus
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Lantus insulin once per day and blood glucose outcomes was studied during the first overnight visit; then the subject was discharged on NPH on twice per day NPH. Upon the second overnight visit, NPH insulin and blood glucose outcomes was studied.
  If the participant entered the study on NPH, NPH insulin given twice per day and blood glucose outcomes was studied during the first overnight visit; then the subject was discharged on once per day Lantus. Upon the second overnight visit, Lantus insulin and blood glucose outcomes was studied
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — BMI (kg/m2) was calculated from measured height and weight. Height was obtained using a wall mounted stadiometer and weight was performed using a digital scale.
  kg/m2 | 25.8 (3.3)
C-peptide [Mean (Standard Deviation); unit: nmole/L] — Fasting blood was drawn. C-peptide (nmole/L) was determined.
  nmole/L | 0.1 (0)
Diabetes duration [Mean (Standard Deviation); unit: years] — Self reported duration of type 1 diabetes.
  years | 22.8 (10.2)
Type of Insulin at First Overnight Visit [Number; unit: participants] — Participants entered the study on either Lantus or NPH. .
  participants
    Lantus (glargine) | 10
    NPH | 5
Fast Acting Insulin [Number; unit: participants]
  Humalog | 8
  Novolog | 6
  Regular | 1

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Area Under the Curve (AUC)
Description: Cumulative sum of repeatedly measured blood glucose values (mg/dl) beginning at 22:00, then hourly till 08:00. Participants were monitored during two overnight sampling periods. One overnight was while the participant was on neutral protamine Hagedorn (NPH) insulin as the long acting insulin; the other overnight was glargine (Lantus) insulin as the the long acting insulin.
Time Frame: Overnight
Population: All participants received either NPH or glargine (Lantus) on separate overnight sampling periods.
Measure: Mean (Standard Deviation); unit: mg*10hr/dL
Groups:
- Glargine (Lantus) Insulin: Glargine (Lantus) was given once per day at 22:00 on the evening of the overnight admission.;
- NPH Insulin: NPH was given at 22:00 on the evening of the overnight admission.
Arm/Group | Glargine (Lantus) Insulin | NPH Insulin
Number analyzed (Participants) | 15 | 15
mg*10hr/dL | 1673.33 (760.7) | 1395 (384.9)
Statistical Analysis 1: Comparison: Glargine (Lantus) Insulin vs NPH Insulin; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; No adjustments were made. T-test type: Paired samples t-test (df=14) was performed using 15 within subject differences; Mean Difference (Final Values) = 277.9, 95% CI 2-sided [-75.9 to 631.6], Standard Error of Mean 164.9 — The comparative measures was defined as (mean AUC of glargine (Lantus)) minus (mean AUC of NPH)

2. Secondary Outcome: Insulin Dose
Description: NPH or glargine (Lantus) was given at 22:00 to provide blood glucose coverage during the overnight hours.
Time Frame: Overnight
Measure: Mean (Standard Deviation); unit: units
Groups:
- Glargine (Lantus) Insulin: Glargine (Lantus) was given once per day at 22:00 on the evening of the overnight admission.
- NPH Insulin: NPH was the given at 22:00 on the evening of the overnight admission.
Arm/Group | Glargine (Lantus) Insulin | NPH Insulin
Number analyzed (Participants) | 15 | 15
units | 20.2 (11.7) | 20.7 (10.0)
Statistical Analysis 1: Comparison: Glargine (Lantus) Insulin vs NPH Insulin; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Cortisol
Description: Mean cortisol nmol/l during NPH or glargine (Lantus) overnight visit. Hourly cortisol was determined from 22:00 to 8:00.
Time Frame: Overnight
Population: Participants completing both overnight visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: nmol/l
Groups:
- Glargine (Lantus): glargine (Lantus) was given once per day at 22:00 on the evening of the overnight admission.
Arm/Group | Glargine (Lantus) | NPH Insulin
Number analyzed (Participants) | 15 | 15
nmol/l | 380.45 (143.48) | 388.61 (122.1)

4. Secondary Outcome: Glucagon
Description: Mean glucagon mcg/l during NPH or glargine (Lantus) overnight visit. Hourly glucagon was determined from 22:00 to 8:00.
Time Frame: Overnight
Population: Participants completing both overnight visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: mcg/l
Groups:
- Glargine (Lantus) Insulin: Glargine (Lantus) was given at 22:00 on the evening of the overnight admission.
Arm/Group | Glargine (Lantus) Insulin | NPH Insulin
Number analyzed (Participants) | 15 | 15
mcg/l | 58.8 (19.0) | 54.3 (19.0)

5. Secondary Outcome: Growth Hormone
Description: Mean growth hormone ug/l during NPH or glargine (Lantus) overnight visit. Hourly growth hormone was determined from 22:00 to 8:00.
Time Frame: Overnight
Population: Participants completing both overnight visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: ug/l
Arm/Group | Glargine (Lantus) Insulin | NPH Insulin
Number analyzed (Participants) | 15 | 15
ug/l | 1.09 (1.61) | 1.27 (2.3)

6. Primary Outcome: Blood Glucose
Description: Average value of repeatedly measured absolute values beginning at 22:00, then hourly till 08:00. Participants were monitored during two overnight sampling periods. One overnight was while the participant was on NPH insulin as the long acting insulin; the other overnight was glargine(Lantus) insulin as the the long acting insulin.
Time Frame: Overnight
Population: All participants received either NPH or glargine (Lantus) on separate overnight sampling periods.
Measure: Mean (Standard Deviation); unit: mmol/l
Groups:
- Glargine (Lantus) Insulin: Glargine (Lantus) was given once per day at 22:00 on the evening of the overnight admission. .
Arm/Group | Glargine (Lantus) Insulin | NPH Insulin
Number analyzed (Participants) | 15 | 15
mmol/l | 9.6 (0.3) | 7.9 (3.7)
Statistical Analysis 1: Comparison: Glargine (Lantus) Insulin vs NPH Insulin; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During active study participation while on either NPH or Lantus insulin. Approximately, 8-12 weeks.
Groups:
- NPH Insulin: Individuals on NPH insuling as long acting insulin.
- Lantus Insulin: Individuals on Lantus insulin as long acting insulin.
Arm/Group | NPH Insulin | Lantus Insulin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Limitation: delayed and slow participant recruitment due to expansive use of insulin pumps and participants unwilling to cross over to alternate insulin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No